CLINICAL TRIAL: NCT04914325
Title: Patient Satisfaction , Marginal Adaptation And Biocompatibility of Milled Biohpp Polyetheretherketone (PEEK) Single Anterior Crowns Veneered With Two Different Techniques.(Randomized Controlled Clinical Trial)
Brief Title: Patient Satisfaction , Marginal Adaptation And Biocompatibility of Milled Biohpp Polyetheretherketone (PEEK) Single Anterior Crowns Veneered With Two Different Techniques.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Salah Mohamed Qasem, principle investegator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 241020
Record Dates: First submitted 2021-05-22; First posted 2021-06-04 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Patient Satisfaction; Gingival Bleeding
MeSH Terms: conditions — Patient Satisfaction; Gingival Hemorrhage | interventions — polyetheretherketone

STUDY DESIGN:
Intervention Model Description: 1. Recording the sulcus depth and gingival condition prior to preparation. 2. Conservative tooth preparation will be prepared after local anesthesia has been given as required. 3. Full coverage preparation will be carried out . 3. After tooth preparation, adequate 2ry Impression using non aqueous elastomeric impression materials and bite registration will be taken. 5. Fabrication of the temporary restoration using composite resin temporary material and cemented using non Eugenol Zinc Oxide temporary cement. 11.a.iii. Fabrication and cementation of restoration: Bio-HPP will be supplied in the form of discs to fabricate crown core by CAD/CAM technology then veneered with two veneering techniques; the CAD/ CAM and the manual technique using the visio.lign system of appropriate shade. The finished Bio HPP crown will be cemented by adhesive resin cement according to manufacturer instruction.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm :copings veneered with CAD/CAM composite resin (Experimental)
  Interventions: Combination Product: peek
- Control arm : copings veneered with manual layering (Active Comparator)
  Interventions: Combination Product: peek

INTERVENTIONS:
Combination Product: peek — After tooth preparation, adequate 2ry Impression using non aqueous elastomeric impression materials and bite registration will be taken. 5. Fabrication of the temporary restoration using composite resin temporary material and cemented using non Eugenol Zinc Oxide temporary cement. 11.a.iii. Fabrication and cementation of restoration: Bio-HPP will be supplied in the form of discs to fabricate crown core by CAD/CAM technology then veneered with two veneering techniques; the CAD/ CAM and the manual technique using the visio.lign system of appropriate shade. The finished Bio HPP crown will be cemented by adhesive resin cement according to manufacturer instruction

SUMMARY:
Research question For patients in a need for anterior crown, does the use of Milled BioHPP PEEK copings veneered with CAD/CAM composite resin offer better patient satisfaction, marginal adaptation and biocompatibility when compared Milled BioHPP PEEK copings veneered with manual layering? Statement of the problem PEEK exhibits a unique modulus of elasticity close to human bone/dentine so it acts as a shock absorber with stress reducing effect. Moreover from a biologic point of view, PEEK is highly compatible with surrounding tissues and it has very promising surface properties . The use of peek in anterior area is limited due to its opaque nature and grayish color, this drawback has been overcome by the use of composite layering material . PEEK restorations can be veneered with manual or CAD/CAM techniques. Information is lacking regarding the influence of the veneering technique on the patient satisfaction , precision of fit and biocompatibility of these restorations which will in turn influence their performance in patient's satisfaction.

Rationale To achieve high esthetics when using PEEK it must be veneered by esthetic material 3 . It is available to be used manually or to be milled by CAD/CAM. The manual veneering of the PEEK coping with composite might affect the marginal integrity and the surrounding gingival tissues leading to decrease in the patient satisfaction, while the CAD/CAM veneering technique is proposed to have better patient satisfaction , marginal adaptation and an excellent biocompatible effect on the surrounding tissue. The importance of this trial lies in providing an alternative solution to the manual veneering technique, which will, in-turn, provide better restoration longevity results

Aim of the study:

The aim of this study is to evaluate the patient satisfaction ,marginal adaptation and biocompatibility of milled BioHPP PEEK copings veneered with CAD/CAM composite resin and compare them to milled BioHPP PEEK copings veneered with manual layering.

Null hypothesis:

There is no difference in the patient satisfaction, marginal adaptation and biocompatibility between milled BioHPP PEEK copings veneered with CAD/CAM composite resin and milled BioHPP PEEK copings veneered with manual layering.

Primary objective: - The Primary outcome: : patient satisfaction of the two groups will be assessed by rating score 0 unaccepted , 1 good , 2 excellent - Secondary outcome: Marginal adaptation of the two groups will be assessed using the modified Ryge criteria. - Tertiary outcome: Biocompatibility (Bleeding). Signs of inflammation and bleeding of the two groups will be recorded after clinical examination and probing using periodontal probe Trial design: - Randomized clinical trial

Eligibility criteria:

Inclusion criteria:

All subjects are required to be: 1-From 18-50 years old, be able to read and sign the informed consent document. 2- Have no active periodontal or pulpal diseases, have teeth with good restorations 3- Psychologically and physically able to withstand conventional dental procedures 4- Patients in a need for anterior crown. 5- Able to return for follow-up examinations and evaluation Exclusion criteria

1. Patient less than 18 or more than 50 years 2. Patient with active resistant periodontal diseases 3. Patients with poor oral hygiene and uncooperative patients 4. Pregnant women 5. Patients in the growth stage with partially erupted teeth 6. Psychiatric problems or unrealistic expectations

DETAILED DESCRIPTION:
Intervention: Examination and diagnosis: - Selection and examination of the patients according to inclusion and exclusion criteria. Diagnosis of the patients' chief complaint and teeth that will be involved in this study will be done then performing proper scaling and polishing procedure, Primary impression will be taken to produce study cast. The patients will be asked to maintain good oral hygiene measures by using tooth brush twice daily. - Taking a pre-operative professional photo, Tooth preparation procedure: Recording the sulcus depth and gingival condition prior to preparation, Conservative tooth preparation will be prepared after local anesthesia has been given as required., Full coverage preparation will be carried out , After tooth preparation, adequate 2ry Impression using non aqueous elastomeric impression materials and bite registration will be taken., Fabrication of the temporary restoration using composite resin temporary material and cemented using non Eugenol Zinc Oxide temporary cement, Fabrication and cementation of restoration: Bio-HPP will be supplied in the form of discs to fabricate crown core by CAD/CAM technology then veneered with two veneering techniques; the CAD/ CAM and the manual technique using the visio.lign system of appropriate shade. The finished Bio HPP crown will be cemented by adhesive resin cement according to manufacturer instruction, Criteria for discontinuing: Restoration will be removed when there are any signs of leakage, fracture or severe post-operative pain due to pulpal response and replaced by a temporary restoration cemented with Ca (OH) cement in order to alleviate pain, Strategies to improve adherence to intervention protocol: - ''In the first visit, a Face to Face adherence session will be held in which the patient should be informed about the study steps and how to maintain oral hygiene measures. Further sessions will occur at the follow-up visits.8 Participant patients will be asked about any problems they are having. Patients will be recalled every three months for one year for follow up visits. Permitted or prohibited interventions: Oral hygiene measures are permitted for enhanced results while using hard tooth brushes or abrasive containing tooth paste after intervention are prohibited.

ELIGIBILITY:
Inclusion Criteria:

All subjects are required to be:

1. From 18-50 years old, be able to read and sign the informed consent document.
2. Have no active periodontal or pulpal diseases, have teeth with good restorations
3. Psychologically and physically able to withstand conventional dental procedures
4. Patients in a need for anterior crown.
5. Able to return for follow-up examinations and evaluation -

Exclusion Criteria:

1. Patient less than 18 or more than 50 years
2. Patient with active resistant periodontal diseases
3. Patients with poor oral hygiene and uncooperative patients
4. Pregnant women
5. Patients in the growth stage with partially erupted teeth
6. Psychiatric problems or unrealistic expectations -

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2023-01-22 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
patient satisfaction of the two groups will be assessed | one year
  rating score 0 unaccepted , 1 good , 2 excellent

SECONDARY OUTCOMES:
Marginal adaptation of the two groups will be assessed u | one year
  using the modified Ryge criteria/- Alpha (A) No visible evidences of crevice along the margins; no catch or penetration of the explorer.
  * Bravo (B) Visible evidence of crevice and/or catch of explorer; no penetration of the explorer.
  * Charlie (C) Visible evidence of crevice and penetration of the explorer

OTHER OUTCOMES:
Biocompatibility (Bleeding) | one year
  Signs of inflammation and bleeding of the two groups will be recorded after clinical examination using periodontal probe

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Salah, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Visit 1: Preoperative records, face-to-face adherence reminder session, clinical, radiographic examination, intraoral photographs and primary impression for diagnostic cast construction. Visit 2: Teeth preparation, secondary impression using addition silicone rubber base material† and temporary restoration. Visit 3: placement and temporary cementation of the interim restoration using temporary cement.
  Visit 4: try in of the coping. Visit 5: placement of final restoration Evaluation of the restoration immediately and follow up visit at (T0, T6, T12)